CLINICAL TRIAL: NCT03819322
Title: Transplantation of Livers of Hepatitis C (HCV) Seropositive Donors to HCV Seronegative Recipients With Subsequent Therapy With Sofosbuvir/Velpatasvir (Epclusa®)
Brief Title: The Use of Hepatitis C Positive Livers in Hepatitis C Negative Liver Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fernanda P Silveira, MD, MS (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor-Investigator, Fernanda P Silveira, MD, MS, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100082
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Liver Transplant; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCV seropositive non-viremic (HCV Ab+/NAT-) donor (Experimental): Liver recipients will be monitored for HCV for one year following transplant. When HCV RNA is detected, the transmission-triggered treatment phase will be initiated.
  Recipients will be treated with 12-week oral course of sofosbuvir/velpatasvir (Epclusa®), a fixed-dose combination of a nucleotide analogue HCV NS5B polymerase inhibitor (sofosbuvir - 400mg) and a NS5A inhibitor (velpatasvir - 100mg).
  Interventions: Drug: sofosbuvir/velpatasvir
- HCV seropositive viremic (HCV Ab+/NAT+) donor (Experimental): Post-operative day 1, liver recipients will be treated with 12-week oral course of sofosbuvir/ velpatasvir (Epclusa®), a fixed-dose combination of a nucleotide analogue HCV NS5B polymerase inhibitor (sofosbuvir - 400mg) and a NS5A inhibitor (velpatasvir - 100mg).
  Interventions: Drug: sofosbuvir/velpatasvir

INTERVENTIONS:
Drug: sofosbuvir/velpatasvir — 12 week, oral, fixed dose
  Other Names: Epclusa

SUMMARY:
This is an open-label, pilot trial to test the safety and efficacy of transplantation of livers from Hepatitis C seropositive non-viremic (HCV Ab+/NAT-) and HCV seropositive viremic (HCV Ab+/NAT+) donors to HCV seronegative recipients on the liver transplant waitlist. Treatment and prophylaxis will be administered, using a transmission-triggered approach for the first scenario (HCV Ab+/NAT- donors, arm 1) and a prophylaxis approach for the later scenario (HCV Ab+/NAT+ donors, arm 2).

DETAILED DESCRIPTION:
This is a prospective, single center, pilot, open-label study of transplantation of livers of HCVAb+ donors to HCVAb- recipients with subsequent therapy with sofosbuvir/velpatasvir (Epclusa®). Recipients of a liver from HCVAb+/NAT- donors will be in arm 1 (the transmission-triggered arm) of the study. In this arm, the study will monitor transmission of HCV by measuring HCV RNA in liver transplant recipients. If HCV RNA is detected, indicating transmission of HCV, recipients will be treated with sofosbuvir/velpatasvir (Epclusa®) for 12 weeks. Virological response will be assessed at 4 weeks, end of treatment and 12 weeks after completion of therapy.

Recipients of a liver from HCVAb+/NAT+ donors will be in arm 2 (the prophylaxis arm) of the study. In this arm, patients will be started on a 12-week course of sofosbuvir/velpatasvir (Epclusa®) immediately post-operatively and will undergo close monitoring of HCV RNA for evidence of transmission.

To be eligible for the study, subjects need to be listed for liver transplantation, be not infected with HCV, HBV or HIV, and sign informed consent.

ELIGIBILITY:
Inclusion criteria (recipients):

1. Patients with end-stage liver disease listed for liver transplantation at UPMC.
2. Age ≥ 18
3. No available living liver donor
4. Listed for an isolated liver transplant at UPMC
5. Have panel reactive antibody level of <98%
6. Able to travel to UPMC for routine post-transplant visits and study visits for a minimum of 12 months after transplantation
7. Able to provide informed consent
8. Be willing to use a contraceptive method for a year after transplant

Exclusion criteria (recipients):

1. HIV positive
2. HCVAb or HCV RNA positive
3. Presence of behavioral risk factors for contracting HCV. These behavioral risk factors are current injection drug use, current intranasal illicit drug use, current percutaneous/parenteral exposures in an unregulated setting.
4. Hepatitis B surface antigen positive
5. History of atrial fibrillation requiring the use of amiodarone over the past 12m
6. Receipt of prior organ transplant
7. Waitlisted for a multi-organ transplant
8. Pregnant women
9. Known allergy to sofosbuvir/velpatasvir
10. Any condition, psychiatric or physical, that in the opinion of the investigator would make it unsafe to proceed with transplantation or interfere with the ability of the subject to participate in the study

Inclusion criteria (donors):

1. HCV antibody positive
2. HCV NAT negative or positive

Exclusion criteria (donors):

1. Confirmed HIV positive (positive HIV-1 antibody, positive HIV-2 antibody, positive p24 antigen and/or positive HIV NAT)
2. Confirmed HBV positive (positive hepatitis B surface antigen and/or HBV NAT)
3. Known ongoing therapy for HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Adverse events | 5 years
  Rate of adverse events due to sofosbuvir/velpatasvir (Epclusa) in study participants in each experimental group
HCV free at 1 year | 1 year
  Proportion of participants in each experimental group who are free of HCV at 1 year following transplantation

SECONDARY OUTCOMES:
Transmission rate of HCV from HCVAb+/NAT- donors to HCVAb- recipients | 5 years
  Transmission rate of HCV from HCVAb+/NAT- donors to HCVAb- recipients
Incidence of allograft rejection | 5 years
  Incidence of allograft rejection at 5 years
Incidence of graft loss | 5 years
  Incidence of graft loss at 5 years
All-cause mortality | 5 years
  All-cause mortality at 5 years
Waitlist time after enrollment | 5 years
  Waitlist time after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Silviera, MD, Study Director — University of Pittsburgh; Naudia Jonassaint, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual patient data outside of our investigative team. Aggregate data will be shared in publications as appropriate.